CLINICAL TRIAL: NCT02148367
Title: Effect of Administration of Recombinant Erythropoietin on Numbers of Circulating Endothelial Progenitor Cells in Patients With Persistent Symptoms During the Subacute Period After TBI
Brief Title: Effect of Recombinant Erythropoietin on Numbers of Circulating Endothelial Progenitor Cells in Subacute TBI
Acronym: TBI-EPO
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Publication of recent trials showing no effect of EPO in TBI.
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ramon Diaz-Arrastia, Professor of Neurology, Uniformed Services University of the Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: T-N-2695; 306135-7.01-60855 (Other Grant/Funding Number: HJF/306135-7.01-60855)
Record Dates: First submitted 2014-05-22; First posted 2014-05-28 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury; Endothelial progenitor cells; Cerebrovascular reactivity; Angiogenesis
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Erythropoietin; Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erythropoietin (EPO) (Active Comparator): Participants (n=20) will receive EPO with a dose of 40,000 IU EPO subcutaneously (s.c.) once weekly for 4 weeks.
  Interventions: Drug: Erythropoietin
- placebo (Placebo Comparator): Participants (n=10) will receive placebo s.c. once weekly for 4 weeks
  Interventions: Drug: Erythropoietin

INTERVENTIONS:
Drug: Erythropoietin — This is a double blind randomized placebo-cotrolled study. Randomization and blinding will be done by the NIH Pharmacy. Participants and study staff will be blinded as to group assignment.Participants randomized into the placebo group will receive placebo once weekly for 4 weeks. In total, 10 participants will be randomized in this group.
  Participants randomized into the experimental group will receive active drug. In total, 20 participants will be randomized in this group. A clinic nurse or physician will administer the study drug, EPO or placebo, to the study participants at the Clinical Center. The study drug is administered by injection under the skin in the arm, leg, or buttock.
  Other Names: Procrit; Epogen

SUMMARY:
* Traumatic brain injury (TBI) is the leading cause of death and disability in people under age 45 in industrialized countries. Significant numbers of US veterans from the wars in Iraq and Afghanistan return with TBI. However, to date, there are no specific neuroprotective treatment options with proven clinical efficacy.
* Erythropoietin (EPO) is approved by the FDA to treat anemia and has comprehensive preclinical data supporting its neuroprotective and neuroregenerative efficacy following traumatic (TBI) and a wide range of other acquired brain insults. Injury to small and medium-sized cerebral blood vessels is a well recognized consequence of TBI. EPO increases production of endothelial progenitor cells (EPCs) and promotes angiogenesis and neovascularization after TBI. EPO also promotes neurogenesis and improves functional recovery in animals after experimental stroke and TBI. Neovascularization is coupled with neurogenesis, and augmentation of both processes by EPO may result in lessened cognitive deficits. Neovascularization by EPO may prevent post-traumatic deficits in cerebrovascular reactivity (CVR), which can be measured noninvasively using magnetic resonance imaging (MRI).
* This proposal is for a randomized, placebo-controlled pilot clinical trial designed to obtain data on the effects of EPO in humans with persistent post-concussive symptoms after TBI. The primary objective is to evaluate effect of 4 week administration of recombinant erythropoietin on numbers of circulating endothelial progenitor cells in patients with persistent symptoms during the subacute period after TBI. This information will guide the design of a future definitive study.

DETAILED DESCRIPTION:
* The study population will include 30 males and females with persistent post-concussive symptoms continuing up to 7 days after TBI. Participants will be military service members or civilians presenting as outpatients for clinical management of TBI or post-concussive symptoms at the Center for Neuroscience and Regenerative Medicine (CNRM)-affiliated hospitals. These include the Walter Reed National Military Medical Center (WRNMMC), Suburban Hospital (SH), and Washington Hospital Center (WHC).
* Design: Participants will be referred to the NIH Clinical Center (CC) from participating hospitals or will be recruited by advertisements through CNRM Recruitment core to receive EPO or placebo. Telephone screening will be carried out to determine tentative eligibility. At the baseline visit, participants will be screened, consented and randomized 2:1 to receive either EPO or placebo with a dose of 40,000 IU EPO subcutaneously (s.c.) (n=20) once weekly for 4 weeks or placebo (n=10). Each participant will have 6 outpatient visits (visits 1-6) performed at the NIH CC. Placebo or active drug will be administered s.c. based on the randomization at visits 1-4; blood will be collected for EPC assays and safety laboratory measurements during each visit. Brain MRI and neuropsychological tests will be performed during visit 1 (before administering EPO or placebo), and visit 5 (one week after final drug administration) and visit 6 (6 months after study enrollment).
* Outcome Measures:
* Primary outcome:

  (1). Effect of 4 weeks of EPO administration on numbers of circulating EPCs in patients with persistent symptoms during the subacute period after TBI (within subject comparison).
* Secondary outcomes:

  (2). Comparison of the change of numbers of circulating EPC's between EPO and placebo groups.

  (3). Effect of 4 weeks of EPO administration on MRI biomarkers of TBI recovery (such as CVR on hypercapnia and global and regional brain volumes by MRI).

  (4). Effect of 4 weeks of EPO administration on plasma biomarkers of angiogenesis and inflammation, such as stem cell factor (SCF), vascular endothelial growth factor (VEGF), stromal-derived factor (SDF-1α); and matrix metalloproteinase-9 (MMP-9).

  (5). Effect of 4 weeks of placebo administration on numbers of circulating EPCs in patients with persistent symptoms during the subacute period after TBI.
* Tertiary outcome:

  (6). Relationship between EPC levels at baseline and after 4 weeks and neuropsychological performance following TBI.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 70 years, inclusive
* History of having sustained a TBI > 3 days and < 7 days prior to enrollment. This evidence will be any one of the following:

  1. GCS 3 - 12 on first presentation to medical attention
  2. Post-traumatic amnesia > 24 hours
  3. TBI-related abnormality on neuroimaging
* Persistent post-concussive symptoms

  1. Three of more of the following symptoms, which started shortly after the trauma and persist for at least up to the time of enrollment:

     * Fatigueability
     * Disordered sleep
     * Headache
     * Vertigo or dizziness
     * Irritability or aggression
     * Anxiety, depression, or affective instability
     * Changes in personality (e.g., social or sexual inappropriateness)
     * Apathy or lack of spontaneity
  2. Symptoms had their onset after trauma, or there is a significant worsening or pre-existing symptoms after trauma.
* Ability to give consent by the participant himself
* Willingness of women of childbearing potential to use effective contraception during this

Exclusion Criteria:

* Contraindication to EPO therapy:

  1. Known allergy to EPO, hypersensitivity to mammalian cell-derived products, or hypersensitivity to albumin
  2. Serum hemoglobin > 16 g/dL in a male patient or > 14 g/dL in a female patient; or a platelet count > 400,000/mm3 or serum hemoglobin < 10 g/dL in either a male or female patient
  3. liver or kidney disease; the former will be operationally defined as a serum bilirubin > 4 mg/dL, alkaline phosphatase (AP) > 250 U/L, aspartate aminotransferase (SGOT, AST) > 150 U/L, alanine aminotransferase (SGPT, ALT) >150 U/L, or Moderately decreased GFR 30-59 ml/min/1.73m2
  4. Pregnancy or lactating; note that a negative pregnancy test will be required if the patient is a female of childbearing potential
* Use of EPO one month prior to the randomization
* Suspicion of a coagulation disorder associated with bleeding (PTT>45 or INR>1.7, spontaneously out of normal range)
* Pre-existing and active major disabling psychiatric disorder (e.g., schizophrenia or bipolar disorder), or other neurological disease (epilepsy, multiple sclerosis, developmental disorder) not related to TBI
* History of heart disease or heart attack, congestive heart failure, stroke, venous thromboembolism.
* History of disorders that predispose to coagulation (e.g. polycythemia vera, essential thrombocytosis, or thrombotic thrombocytopenic purpura).
* Uncontrolled hypertension, defined as above 140/90 mm Hg in three measurements in two separate visits despite antihypertensive therapy.
* Known malignant conditions, e.g., melanoma, breast, brain, lung tumor or prostate cancer
* Terminal medical diagnosis consistent with survival < 1 year
* Planned surgical procedure during duration of the study
* Current use of Coumadin or other blood thinners (e.g. Pradaxa, Heparin, Lovenox).
* Any history of previous deep venous thrombosis (DVT), pulmonary embolization (PE), or other thromboembolic event
* Current participation in other interventional clinical trial
* Current use of iron supplements
* Evidence of penetrating brain injury
* Contraindication to MRI scanning
* No adherence to use of effective method of contraception for females of childbearing potential for time from enrollment to the study until 2 weeks after completion of the study drug

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Effect of 4 weeks of EPO administration on numbers of circulating EPCs in patients with persistent symptoms during the subacute period after TBI (within subject comparison). | Four weeks of treatment
  Study participants (n=20) will receive EPO once weekly 40,000 IU for 4 weeks. Blood will be collected for EPC assays during each visit. EPC numbers determined after the drug administration will be compared to EPC numbers obtained at the baseline visit.

SECONDARY OUTCOMES:
Comparison of the change of numbers of circulating EPC's between EPO and placebo groups. | Four weeks of treatment
  Numbers of EPC in treatment group will be compared numbers of EPC determined in placebo group during four weeks of drug/placebo administration.
Effect of 4 weeks of EPO administration on plasma biomarkers of angiogenesis and inflammation, such as stem cell factor (SCF), vascular endothelial growth factor (VEGF), stromal-derived factor (SDF-1α); and matrix metalloproteinase-9 (MMP-9) | Four weeks of threatment
  Biomarkers of of angiogenesis and inflammation will be evaluated in the treatment and placebo groups.
Effect of 4 weeks of placebo administration on numbers of circulating EPCs in patients with persistent symptoms during the subacute period after TBI. | Four weeks of treatment
  EPC numbers will be studied in TBI participants receiving placebo to elucidate natural history of temporal profiles of EPC after TBI.

OTHER OUTCOMES:
Relationship between EPC levels at baseline and after 4 weeks and neuropsychological performance following TBI. | 5 weeks and 6 months after the TBI
  Neuropsychological performance using subset of Common Data Elements will be studied 5 weeks and 6 months after TBI. These neuropshychological outcomes will be related to levels of EPC on admission and after 4 weeks of the drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Diaz-Arrastia, MD, PhD, Principal Investigator — Uniformed Services University of the Health Sciences; Eric Wassermann, MD, Principal Investigator — National Institutes of Health (NIH)
Locations (1):
- National Institutes of Health, Clinical Center., Bethesda, Maryland, United States

REFERENCES:
- [Background] Bahlmann FH, De Groot K, Spandau JM, Landry AL, Hertel B, Duckert T, Boehm SM, Menne J, Haller H, Fliser D. Erythropoietin regulates endothelial progenitor cells. Blood. 2004 Feb 1;103(3):921-6. doi: 10.1182/blood-2003-04-1284. Epub 2003 Oct 2. PMID 14525788
- [Background] Guo X, Liu L, Zhang M, Bergeron A, Cui Z, Dong JF, Zhang J. Correlation of CD34+ cells with tissue angiogenesis after traumatic brain injury in a rat model. J Neurotrauma. 2009 Aug;26(8):1337-44. doi: 10.1089/neu.2008.0733. PMID 19226208
- [Background] Bogoslovsky T, Chaudhry A, Latour L, Maric D, Luby M, Spatz M, Frank J, Warach S. Endothelial progenitor cells correlate with lesion volume and growth in acute stroke. Neurology. 2010 Dec 7;75(23):2059-62. doi: 10.1212/WNL.0b013e318200d741. PMID 21135380